CLINICAL TRIAL: NCT00430287
Title: Correlation of DDLS Grading to OCT, HRT, and HVF
Brief Title: Does the Optic Disc Grading Done Visually by Your Doctor Agree With Optic Nerve Testing Which is Done by Machines?
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jonathon Myers, Attending Surgeon, Wills Eye
Other Study IDs: 06-775
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Open Angle Glaucoma
Keywords: primary open angle glaucoma; low tension glaucoma; pigmentary glaucoma; exfoliative glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Primary open angle glaucoma: Patients with a form of primary open angle glaucoma
- 2: No known eye disease (controls): Patients with no known eye disease (controls)

SUMMARY:
The purpose of this study is to determine how well the DDLS (Disc Damage Likelihood Scale) (which is a method used by the eye doctor to evaluate how healthy the optic nerve is) measures up to the standard glaucoma tests: OCT (Optical Coherence Tomography), the HRT (Heidelberg Retinal Tomography) and the HVF (Humphrey Visual Field).

DETAILED DESCRIPTION:
The Disc Damage Likelihood Scale (DDLS) has been shown to be a reproducible method for clinicians to evaluate the optic nerve for glaucomatous damage and is highly correlated to diagnosis of glaucoma, severity of glaucoma as evidenced by visual field loss and Heidelberg Retina Tomography (HRT) evaluation. In comparison with the commonly used cup-disc ratio, the DDLS has less inter-observer variation and captures glaucomatous aspects of the optic nerve not assessed by the cup-disc ratio. The optic nerve imagers do not have the potential to completely replace the clinical examination of the optic nerve since they do not assess many critical features such as optic nerve pallor, hemorrhages, asymmetry of disc size, edema, etc. The DDLS presents the opportunity to provide a system to clinicians to increase the quality and objectivity of clinical optic nerve evaluation. The purpose of this study is to investigate the correlation of the DDLS grading to OCT, HRT and HVF testing of glaucomatous and normal optic nerves.

ELIGIBILITY:
Inclusion Criteria:

* Vision 20/50 or better
* Less than 3 diopters of astigmatism
* 3 diopters or less of myopia or hyperopia
* Pattern Standard Deviation on HVF less than 2.5dB in normals
* Pattern Standard Deviation on HVF greater than 2.5 db in glaucoma patients

Exclusion Criteria:

* Abnormalities of cornea or ocular media
* Significant ocular pathologies affecting visual field
* History of hypotony
* Ocular surgery within 6 months
* Nystagmus
* Unreliable visual fields
* OCT signal strength scan less than 6

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: glaucoma service
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Myers, MD, Principal Investigator — Wills Eye Glaucoma Service
Locations (1):
- Wills Eye Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript has been published.